CLINICAL TRIAL: NCT05348590
Title: Nutritional Assessment Project In Surgical Patients Focused On Body Composition And Functionality
Brief Title: Phase-Germ Project: Muscle Mass and Phase Angle in Surgical Patient
Acronym: FASE-GERM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Hospital Universitario Virgen de la Victoria (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jose-M Ramirez, Prof., Universidad de Zaragoza
Other Study IDs: UZaragoza 4
Record Dates: First submitted 2022-04-20; First posted 2022-04-27 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-12

CONDITIONS: Surgery; Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current nutritional diagnostic tools have serious limitations in certain groups of patients such as colon or ovarian cancer with high rates of overweight and obesity in which traditional anthropometric assessment is limited.

The objective of the project is to establish a comprehensive nutritional assessment in surgical patients assessed in intensified recovery programs in Surgery at a national level, including new techniques aimed at measuring muscular and functional affection.

DETAILED DESCRIPTION:
Current nutritional diagnostic tools have serious limitations in certain groups of patients such as colon or ovarian cancer with high rates of overweight and obesity in which traditional anthropometric assessment is limited with underdiagnosis of malnutrition and possible effect on therapeutic toxicity and other complications.

The objective of the project is to establish a comprehensive nutritional assessment in surgical patients assessed in intensified recovery programs in Surgery at a national level, including new techniques aimed at measuring muscular and functional affection in order to make a more precise diagnosis and a better prediction of complications and morbidity and mortality.

In this group of patients with moderate or severe malnutrition, it is important to evaluate new techniques aimed at nutritional assessment with assessment tools focused on the morpho-functional diagnosis of malnutrition.

From a scientific point of view, the following nutritional assessment techniques are being incorporated:

1- BIOIMPEDANCIOMETRY: Non-invasive technique, relatively inexpensive and easily transportable. 2- MUSCLE ULTRASOUND: The application of ultrasound for the morphological and structural study of muscle mass is an emerging technique.

3- DYNAMOMETRY: Dynamometry is one of the 6 criteria that define malnutrition according to ASPEN. It is a very sensitive parameter. 4- FUNCTIONAL TESTS: The execution or performance tests consist of the development of a series of physical activities related to mobility, walking or balance. Their results are related to those of the scales that assess the Activities of Daily Living (IADL).

The main OBJECTIVES of the study are:

1. To establish a record of the prevalence of malnutrition in the surgical area based on morpho-functional techniques (adapted GLIM criteria).
2. To evaluate the implementation of morpho-functional diagnostic tools in said area (Bioimpedanciometry, muscle ultrasound and dynamometry).
3. To correlate the clinical-prognostic aspects with the clinical situation of the patient (morbidity-mortality, adverse effects associated with the disease itself or with the treatment, adaptation of the therapeutic regimen, quality of life...)

Design: Prospective observational study, following the usual clinical practice without altering the flow of visits to clinical nutrition clinics.

Patients: Patients presenting with acute or chronic disease-related protein calorie malnutrition on outpatient follow-up treatment by a multimodal salvage surgery program.

Variables:

* Assessment of Nutritional Status:

  * Global Subjective Assessment (GSV) Questionnaire: ANNEX 2
  * Current weight (measured or estimated), usual weight, weight for calculations (adjusted weight in obese, weight without edema in malnourished), height (measured or estimated), BMI (measured or estimated), arm circumference.
  * Electrical bioimpedance measurement (model (50khz) Akern BIA 101): The following data will be obtained: TBW (total body water, L), ECW (extracellular water, L), ICW (intracellular water, L), FFM (lean mass, Kg ), FM (fat mass, Kg), BCM (cell mass, Kg), ASMM (appendicular muscle mass, Kg), SMI (muscle mass index, Kg), Hydration %.
  * Electrical bioimpedance measurement (TANITA Model TBF-300): Fat mass, in percent, Lean mass, in kilograms, Total body water, in percent, Body mass index, basal metabolism.
  * Abdominal and muscle ultrasound (mindray z6 probe 7l4p):

    * Abdominal echo: total, superficial and pre-peritoneal adipose tissue. Muscle echo (measured in centimeters).
    * Muscle echo: Area, circumference, axes and adipose tissue (measured in centimeters)
* Analytical parameters: A blood test will be requested which will include the following determinations:

  * Total cholesterol and triglycerides, in milligrams per deciliter.
  * C-reactive protein, in milligrams per deciliter.
  * Albumin, in grams per deciliter.
  * Prealbumin, in milligrams per deciliter.
  * Lymphocytes, in microliters,
* Functional parameters:

  * Get Up and Go Test: "get up and go" test: The patient sits on a chair, tells him to get up (start of test and timing), walks 3 meters and sits back on the initial chair (end of timing). ). Interpretation: < 20 seconds: normal, > 20 seconds: increased risk of falling.
  * Jamar® type dynamometers are the most widely used in international studies and have various grip positions. Make 3 measurements with their subsequent average, measured in Kilograms.

Data collection and analysis: Record of described variables were be included in an "on line"database available to all centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old, scheduled for major abdominal surgical surgery, due to malignant or benign causes.

Exclusion Criteria:

* Urgent Surgery. Patients ASA (American Society of Anesthesiology) IV or higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, scheduled for major abdominal surgical surgery, due to malignant or benign causes (It is defined as complex major surgery that lasts more than two hours or it is estimated that it may require the transfusion of at least 2 red cell concentrates or it is estimated a loss greater than or equal to 15% of the patient's blood volumen)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with malnutrition | 1 month perioperatory
  Number of patient operated on with malnutrition
To asses the value of Morphofunctional tools in detect malnutrition | 1 month
  Accuracy of morphofunctional test in diagnosing malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Ramirez, Study Director — Universidad de Zaragoza
Locations (1):
- Hospital Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sjoblom B, Gronberg BH, Benth JS, Baracos VE, Flotten O, Hjermstad MJ, Aass N, Jordhoy M. Low muscle mass is associated with chemotherapy-induced haematological toxicity in advanced non-small cell lung cancer. Lung Cancer. 2015 Oct;90(1):85-91. doi: 10.1016/j.lungcan.2015.07.001. Epub 2015 Jul 9. PMID 26198373
- [Background] Garcia Almeida JM, Garcia Garcia C, Vegas Aguilar IM, Bellido Castaneda V, Bellido Guerrero D. Morphofunctional assessment of patient s nutritional status: a global approach. Nutr Hosp. 2021 Jun 10;38(3):592-600. doi: 10.20960/nh.03378. PMID 33749304
- [Background] Norman K, Stobaus N, Pirlich M, Bosy-Westphal A. Bioelectrical phase angle and impedance vector analysis--clinical relevance and applicability of impedance parameters. Clin Nutr. 2012 Dec;31(6):854-61. doi: 10.1016/j.clnu.2012.05.008. Epub 2012 Jun 12. PMID 22698802
- [Background] Grundmann O, Yoon SL, Williams JJ. The value of bioelectrical impedance analysis and phase angle in the evaluation of malnutrition and quality of life in cancer patients--a comprehensive review. Eur J Clin Nutr. 2015 Dec;69(12):1290-7. doi: 10.1038/ejcn.2015.126. Epub 2015 Jul 29. PMID 26220573
- [Background] Lukaski HC, Kyle UG, Kondrup J. Assessment of adult malnutrition and prognosis with bioelectrical impedance analysis: phase angle and impedance ratio. Curr Opin Clin Nutr Metab Care. 2017 Sep;20(5):330-339. doi: 10.1097/MCO.0000000000000387. PMID 28548972
- [Background] Paiva SI, Borges LR, Halpern-Silveira D, Assuncao MC, Barros AJ, Gonzalez MC. Standardized phase angle from bioelectrical impedance analysis as prognostic factor for survival in patients with cancer. Support Care Cancer. 2010 Feb;19(2):187-92. doi: 10.1007/s00520-009-0798-9. Epub 2009 Dec 29. PMID 20039074
- [Background] Nunez M, Nunez E, Moreno JM, Segura V, Lozano L, Maurits NM, Segur JM, Sastre S. Quadriceps muscle characteristics and subcutaneous fat assessed by ultrasound and relationship with function in patients with knee osteoarthritis awaiting knee arthroplasty. J Clin Orthop Trauma. 2019 Jan-Feb;10(1):102-106. doi: 10.1016/j.jcot.2017.11.014. Epub 2017 Nov 24. PMID 30705541
- [Background] Barata AT, Santos C, Cravo M, Vinhas MD, Morais C, Carolino E, Mendes L, Roldao Vieira J, Fonseca J. Handgrip Dynamometry and Patient-Generated Subjective Global Assessment in Patients with Nonresectable Lung Cancer. Nutr Cancer. 2017 Jan;69(1):154-158. doi: 10.1080/01635581.2017.1250923. Epub 2016 Dec 5. PMID 27918868
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- See also: Web of the Spanish Group on MUltimodal Rehabilitation — http://grupogerm.es